CLINICAL TRIAL: NCT04818502
Title: Real World Study of the Tendyne™ Mitral Valve System to Treat Mitral Regurgitation (RESOLVE-MR) (Tendyne™ PMCF Study)
Brief Title: Real World Study of the Tendyne™ Mitral Valve System to Treat Mitral Regurgitation
Acronym: RESOLVE-MR
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10313
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Mitral Valve Regurgitation
Keywords: Tendyne; Tendyne Mitral Valve System; Transcatheter; Mitral Regurgitation; Heart Valve disease; Mitral Valve Regurgitation; Mitral Insufficiency; Transcatheter intervention; Transcatheter Mitral Valve Implantation; Transcatheter Mitral Valve Replacement; Transapical Transcatheter Mitral Valve Implantation
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tendyne™ Mitral Valve System — Transcatheter mitral valve implantation (TMVI) using the Tendyne™ Mitral Valve System , in which a bioprosthetic valve is implanted within the native mitral valve.
  Other Names: Transcatheter Mitral Valve Implantation (TMVI)

SUMMARY:
To evaluate the safety and performance of the Tendyne™ Mitral Valve System when used as intended in a contemporary, real-world setting.

DETAILED DESCRIPTION:
The Tendyne RESOLVE-MR study (Real World Study of the Tendyne™ Mitral Valve System to Treat Mitral Regurgitation) is a prospective, single arm, multi-center, PMCF study, which will be used to support the CE Mark requirement of monitoring safety and performance for any complications or issues arising in a post-market setting.

The objective of the Tendyne RESOLVE-MR study is to confirm the safety and performance of the Tendyne Mitral Valve System in patients with symptomatic, moderate-to-severe or severe mitral regurgitation (MR) who are considered by the local heart team as eligible for a transapical transcatheter mitral valve implantation in a real-world setting. This clinical study is intended to satisfy post-market clinical follow-up requirements of CE Mark.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is indicated for the Tendyne Mitral Valve System per the Instructions for Use.
2. Patient is willing and able to comply with all follow-up requirements through five years, including study-required testing, medications, and attending all follow-up visits.
3. Patient provides written informed consent prior to any study-specific procedure.

Exclusion Criteria:

1. Patient is in another clinical study that may impact the follow-up or results of this study.
2. Patient is pregnant or nursing or plan to become pregnant during the study follow-up period.
3. Patient is under the age of 18 or age of legal consent.
4. Patient has other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, may limit the subject's ability to participate in the clinical study or to comply with follow-up requirements.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects of all genders from the population of patients meeting indications for a Tendyne implant as stated within the IFU. Subjects must meet all eligibility criteria and provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint for MR Elimination at 1 Year | At 1 year
  The primary endpoint MR Elimination will be assessed at one year post-procedure and is defined as original Tendyne valve remains implanted, free from surgical removal/replacement or transcatheter mitral valve implantation (valve-in-valve), and MR < Grade I (mild, measured by Echocardiographic Core Lab)

SECONDARY OUTCOMES:
Procedure Safety (PS) | Day 0, at exit procedure room
  This will be assessed at exit from the procedure room and is defined as freedom from procedural mortality, unplanned surgical or interventional procedures related to the Tendyne valve or access procedure.
Freedom from LVOT Obstruction (LVOTO) at 30 Days | At Day 30
  This will be assessed at 30 days post-procedure and is defined as mean LVOT gradient increase <10 mmHg from baseline (measured by the Echo Core Lab), and free of unplanned intervention for LVOTO.
Freedom from Paravalvular Leak (PVL) at 30 Days | At Day 30
  This will be assessed at 30 days post-procedure and is defined as the Tendyne prosthesis PVL ≤ mild (Grade I), as measured by the Echo Core Lab.
Left Ventricle Reverse Remodeling at 1 Year | At 1 Year
  This will be assessed at 1-year post-procedure and is defined as the proportion of survivors at one year with baseline Left Ventricle End Diastolic Volume Index (LVEDVi) > 96ml/m2 that experience 10% or greater reduction in LVEDVi at one year (assessed by the Echo Core lab).
All-Cause Mortality at 30 Days | At Day 30
  This will be assessed at 30 days post-procedure and is defined as the proportion of subjects who die within 30 days post-procedure for any cause.
Long-term Device Durability (LDD) at 5 Years | At 5 Years
  This will be assessed at 5 years post-procedure and is defined as original Tendyne device remains implanted, free from surgical removal/replacement or transcatheter mitral valve implantation (valve-in-valve), and free from Structural Valve Dysfunction

CONTACTS AND LOCATIONS:
Locations (36):
- Kepler University Hospital, Linz, Austria
- UZ Gasthuisberg, Leuven, Belgium
- Czechia (3):
  - University Hospital Olomouc, Olomouc
  - IKEM Prague, Prague
  - Hospital AGEL Trinec-Podlesi, Třinec
- France (5):
  - Bordeaux University Hospital, Bordeaux
  - CHRU de Lille, Lille
  - Lyon University Hospital, Lyon
  - Rennes University Hospital, Rennes
  - Clinique Pasteur, Toulouse
- Germany (12):
  - Heart and Diabetes Center NRW, Bad Oeynhausen
  - German Heart Center Berlin, Berlin
  - University Hospital Bonn, Bonn
  - Universitätsclinic Cologne, Cologne
  - University Hospital Frankfurt, Frankfurt
  - University Heart Center Hamburg, Hamburg
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Leipzig Heart Center, Leipzig
  - University Medical Center Mainz, Mainz
  - German Heart Center Munich, Munich
  - Ludwig-Maximilians-Universität (LMU) München / Campus Großhadern, München
  - Robert-Bosch Krankenhaus, Stuttgart
- Israel (2):
  - Shaare Zedek Jerusalem, Jerusalem
  - Sheba Medical Centre, Tel Aviv
- Italy (3):
  - Lancisi Cardiovascular Center - Politechnic University of Marcher, Ancona
  - AOU Civili Brescia, Brescia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- MUMC+, Maastricht, Netherlands
- Oslo University Hospital, Oslo, Norway
- Saudi Arabia (3):
  - King Fahad Armed Forces, Jeddah
  - King Fahad Medical City, Riyadh
  - King Faisal Specialist Hospital & Research Center, Riyadh
- Clinico San Carlos, Madrid, Spain
- Switzerland (2):
  - University Hospital Basel, Clinic for Cardiac Surgery, Basel
  - Insel Bern, Bern
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No